CLINICAL TRIAL: NCT05850182
Title: A Pilot Study to Investigate the Effects of Lifestyle Intervention on Physical Activity and Diet in Patients With Metastatic Prostate Cancer Receiving Novel Hormonal Agents: the ACTIDIET-PRO Study
Brief Title: Lifestyle Intervention in Patients With Metastatic Prostate Cancer
Acronym: ACTIDIET-PRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oncology Institute of Southern Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACTIDIET-PRO
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm treated with lifestyle intervention (Experimental): Patients with prostate cancer will receive a lifestyle intervention on diet and physical activity.
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — 12-week lifestyle intervention including adherence to a personalized balanced dietary regimen (low total fat, low saturated fat, high ω3 fatty acids, optimized protein content, low simple sugars) combined with regular physical activity (including physiotherapy sessions and self-training).

SUMMARY:
The proposed pilot study aims at determining the feasibility of a lifestyle intervention including adherence to a personalised dietary regimen combined with regular physical activity in patients newly diagnosed with prostate cancer under androgen deprivation therapy.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is among the most frequent tumor types and is the second deadliest type of cancer in men.

PCa has a multifactorial aetiology; modifiable environmental factors, including diet and obesity, have been associated with prostate carcinogenesis. Furthermore, patients with PCa are treated with androgen deprivation therapy (ADT), which has negative effects on the cardiovascular system and body composition, particularly on the fat and muscle mass, bone health and psychological wellbeing.

Data in the current literature suggests that a lifestyle intervention e.g. with targeted and supervised exercise therapy or a dietary intervention with a prudent dietary patternmay positively influence the quality of life and the course of the disease of patients under ADT. However, conclusive data is missing.

The proposed pilot study aims at determining the feasibility and the effect of a lifestyle intervention including adherence to a personalised dietary regimen combined with regular physical activity in patients newly diagnosed with PCa under ADT.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration.
* Age ≥ 18 years
* Histology of adenocarcinoma of the prostate
* Patients with PCa receiving ADT alone or ADT+NHT (abiraterone, enzalutamide, apalutamide or darolutamide)
* Rising PSA (two consecutively rising PSA levels > 25% above nadir at least three weeks apart), with no evidence of clinical or radiographic progression on instrumental evaluation
* PSA doubling time > 8 weeks
* Continuation of ongoing systemic treatment is deemed feasible by treating physician

Exclusion Criteria:

* Ongoing treatment with docetaxel, cabazitaxel, radionuclides or investigational treatments
* Evidence of clinical progression or progression of disease on imaging
* Bone metastases excluding the safety of physical exercise
* Prior confirmed severe osteoporosis or other diseases affecting the bone with history of fractures
* Clinically significant cardiovascular disease (i.e. myocardial infarction within 6 months before screening; uncontrolled angina within 3 months before screening; congestive heart failure New York Heart Association class 3 or 4; history of clinically significant arrhythmias; uncontrolled hypertension indicated by systolic blood pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg at screening)
* Clinically significant chronic obstructive pulmonary disease
* Any concurrent disease or comorbid condition that interferes with the ability of the patient to participate in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient initiation rate | 12 weeks
  Study initiation rate (total number of patients enrolled divided by the number of patients screened for the study)
Patient retention rate | 12 weeks
  Retention rate (number of patients completing the study divided by total number of patients enrolled at baseline)
Adherence to prescribed training program | 12 weeks
  Adherence rate (fraction of scheduled physical activity appointments/selftrainings attended/carried out by the patients)
Adherence to prescribed dietary regimen | 12 weeks
  Adherence rate (fraction of days of adherence to the prescribed dietary regimen)

SECONDARY OUTCOMES:
Effect of lifestyle intervention on PSA progression | 24 weeks
  Percentage of PSA non-progressors (patients with <25% PSA rise compared to baseline) at weeks 8, 12 and 24
Effect of lifestyle intervention on PSA levels | 24 weeks
  PSA doubling time calculated with the formula PSA doubling time = ln (2) / PSA Slope [PSA Slope = (ln (PSA level 2) - ln (PSA level 1)) / Time (no. of months)]
Effect of lifestyle intervention on radiographic progression | 24 weeks
  Percentage of patients being free of radiographic progression according to PCWG3 at weeks 12 and 24
Effect of lifestyle intervention on patient-reported quality of life | 24 weeks
  Change in patient-reported quality of life from baseline using Functional Assessment of Cancer Therapy - Prostate (FACT-P) scoring from baseline to weeks 8, 12 and 24
Effect of lifestyle intervention on patient-reported fatigue | 24 weeks
  Change in patient-reported fatigue from baseline using FACIT Fatigue scoring from baseline to weeks 8, 12 and 24
Effect of lifestyle intervention on time to subsequent treatment | 24 months
  Time to a subsequent line of treatment (in weeks)
Effect of lifestyle intervention on plasma lipid signature | 8 weeks
  Concentration of individual lipid types in the plasma of participating patients, change compared to baseline
Effect of lifestyle intervention on plasma immune signature | 8 weeks
  Concentration of inflammatory cytokines in the plasma of participating patients, change compared to baseline
Effect of lifestyle intervention on microbiome composition | 8 weeks
  Differences in community diversity and/or abundance of specific bacterial taxa within the intestinal microbiome prior to or during the lifestyle intervention.
Effect of lifestyle intervention on anthropometric variables | 24 weeks
  Measurement of patient height and body weight and calculation of body-mass index (BMI) at baseline, during and after the lifesyle intervention.
Effect of lifestyle intervention on lean body mass | 12 weeks
  Measurement of the percentage of lean body mass by bioelectrical impedance vector analysis and by magnetic resonance imaging.
Effect of lifestyle intervention on fat body mass | 12 weeks
  Measurement of the percentage of fat body mass by bioelectrical impedance vector analysis and by magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided